CLINICAL TRIAL: NCT00002934
Title: Local Excision Alone for Selected Patients With DCIS of the Breast
Brief Title: Evaluation of Breast Cancer Recurrence Rates Following Surgery in Women With Ductal Carcinoma In Situ
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated when the accrual goal for the low/intermediate grade stratum was reached. The high grade stratum was closed due to slow accrual.
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000065370; U10CA021115 (NIH); E-5194
Record Dates: First submitted 1999-11-01; First posted 2003-04-16 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
Keywords: breast cancer in situ; ductal breast carcinoma
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ; Carcinoma, Ductal, Breast

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pathology Review, Observation and Follow-up (No Intervention): Pathology review, observation and follow-up
  Interventions: Procedure: long-term screening

INTERVENTIONS:
Procedure: long-term screening

SUMMARY:
RATIONALE: The evaluation of breast cancer recurrence rates may improve the ability to plan cancer treatment for patients with breast cancer.

PURPOSE: Study to evaluate the rate of recurrence of breast cancer in women who have had surgery for ductal carcinoma in situ.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate actuarial local in situ and invasive recurrence rates at 5 and 10 years after local excision in women with a favorable ductal carcinoma in situ (DCIS) prognosis.
* Evaluate concordance between institutional pathologists and central review pathologists with respect to diagnosis and grading of DCIS.
* Identify parameters that indicate increased or decreased risk of recurrence in the absence of irradiation.
* Evaluate patterns of salvage of recurrence and rates of breast conservation.
* Evaluate actuarial relapse-free, overall, and cause-specific survival at 5 and 10 years post DCIS excision.

OUTLINE: This is a registration study stratified by histologic grade (high vs low or intermediate) and adjuvant tamoxifen therapy (yes vs no).

Patients receive standard clinical and mammographic follow-up for greater than 10 years. If recurrence occurs, treatment will be at the discretion of the investigators. Patients may receive adjuvant oral tamoxifen daily for 5 years after local excision.

A follow up magnification view mammogram must be taken after the last local excision, and microcalcification must be negative.

Patients are followed every 6 months for the first 10 years, and then annually thereafter.

PROJECTED ACCRUAL: 1000 (500 per stratum) eligible and evaluable patients will be enrolled at an estimated accrual rate of 250 patients per year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven low or intermediate grade ductal carcinoma in situ (DCIS) of the breast

  * No greater than 2.5 cm in the greatest dimension
* OR
* Histologically proven high-grade DCIS of the breast

  * No greater than 1 cm in greatest dimension
* Region of DCIS must be at least 2.5 mm in greatest dimension (mammographic estimate of size allowed where pathologic measurement is impossible)
* DCIS must be non-palpable; detected by a mammogram or found incidentally by a breast biopsy
* Pathologically confirmed negative margins of at least 3 mm
* Breast must be suitable for breast conserving therapy

  * Proper tumor size versus breast size
  * No carcinoma or suspicious mammogram findings in other breast sites
* No prior in situ or invasive breast cancer
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Female

Menopausal status:

* Not specified

Performance status:

* Not specified

Life expectancy:

* Greater than 5 years

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Cardiovascular:

* Not specified

Other:

* No other invasive malignancies within the past 10 years except nonmelanomatous skin cancer or carcinoma in situ of the cervix
* No known HIV infection
* No Paget's nipple disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Not specified

Endocrine therapy:

* Adjuvant tamoxifen allowed

Radiotherapy:

* No prior radiotherapy to breast
* No adjuvant radiotherapy

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 711 (Actual)
Dates: Start 1997-06-25 (Actual); Primary Completion 2007-12 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Actuarial local recurrence rate | Assessed at 5 years
  Rate of in situ or invasive local breast cancer recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Lorie L. Hughes, MD, Study Chair — Emory University
Locations (30):
- United States (29):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center - Indianapolis (Roudebush), Indianapolis, Indiana
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Ireland Cancer Center, Cleveland, Ohio
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Veterans Affairs Medical Center - Tennessee Valley Healthcare System - Nashville Campus, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - CCOP - Green Bay, Green Bay, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee (Zablocki), Milwaukee, Wisconsin
- Pretoria Academic Hospitals, Pretoria, South Africa

REFERENCES:
- [Result] Hughes LL, Wang M, Page DL, Gray R, Solin LJ, Davidson NE, Lowen MA, Ingle JN, Recht A, Wood WC. Local excision alone without irradiation for ductal carcinoma in situ of the breast: a trial of the Eastern Cooperative Oncology Group. J Clin Oncol. 2009 Nov 10;27(32):5319-24. doi: 10.1200/JCO.2009.21.8560. Epub 2009 Oct 13. PMID 19826126
- [Result] Hughes L, Wang M, Page D, et al.: Five year results of intergroup study E5194: local excision alone (without radiation treatment) for selected patients with ductal carcinoma in situ (DCIS). [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-29, S15, 2006.
- [Derived] Solin LJ, Gray R, Hughes LL, Wood WC, Lowen MA, Badve SS, Baehner FL, Ingle JN, Perez EA, Recht A, Sparano JA, Davidson NE. Surgical Excision Without Radiation for Ductal Carcinoma in Situ of the Breast: 12-Year Results From the ECOG-ACRIN E5194 Study. J Clin Oncol. 2015 Nov 20;33(33):3938-44. doi: 10.1200/JCO.2015.60.8588. Epub 2015 Sep 14. PMID 26371148